CLINICAL TRIAL: NCT01648855
Title: Consequences of Circulating Antiangiogenic Factors Involved in Preeclampsia on Intra-uterine Growth Restricted Preterm Newborn
Brief Title: Consequences of Antiangiogenic Factors Involved in Preeclampsia on Intra-uterine Growth Restricted Preterm Newborn
Acronym: ANGIODYS
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI 11030
Record Dates: First submitted 2012-07-20; First posted 2012-07-24 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-06

CONDITIONS: Preterm Birth; Intra-uterine Growth Restriction; Maternal Preeclampsia; Bronchopulmonary Dysplasia
Keywords: Circulating antiangiogenic factors; Preeclampsia; Developing lung; Bronchopulmonary dysplasia
MeSH Terms: conditions — Premature Birth; Bronchopulmonary Dysplasia; Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Preterm babies: Intra uterine growth restricted preterm babies born before 30 weeks of gestational age from mother with preeclampsia
  Interventions: Other: Biological samples

INTERVENTIONS:
Other: Biological samples — To measure the levels of sFlt1, angiogenic and antiangiogenic factors at birth in maternal blood, umbilical cord blood and in the amniotic fluid

SUMMARY:
Preeclampsia complicates about 2-7% of pregnancies and is a major contributor to maternal and neonatal morbidity and mortality worldwide. Imbalance between circulating angiogenic and antiangiogenic factors has emerged as a potential key pathway in the pathophysiology of preeclampsia. Patients with preeclampsia have a higher circulating concentration of antiangiogenic factors (ie, soluble vascular endothelial growth factor receptor-1 [sVEGFR- 1], also called soluble fms-like tyrosine kinase 1 [sFlt1]) and soluble endoglin (sEng)] and a lower maternal circulating concentration of free angiogenic factors (ie, vascular endothelial growth factor [VEGF] and placental growth factor [PlGF]) than patients with a normal pregnancy. Bronchopulmonary dysplasia is the main respiratory sequelae of preterm birth. Its rate increased in preterm infants born from mother with preeclampsia. Recent studies showed that bronchopulmonary dysplasia is consistently accompanied by a reduction in the number of small arteries and on abnormal distribution of vessels within the distal lungs. This is associated with reduced lung VEGF expression. The main objective of this population-based study, ie in intra uterine growth restricted preterm babies born before 30 weeks of gestational age, was to examine whether levels of sFlt1 at birth in maternal and umbilical cord blood and in the amniotic fluid is associated with an increased risk of BPD.

DETAILED DESCRIPTION:
Preeclampsia complicates about 2-7% of pregnancies and is a major contributor to maternal and neonatal morbidity and mortality worldwide. Preeclampsia is the main cause of intra-uterine growth restriction and could lead to a preterm delivery for fetal or maternal indication. Imbalance between circulating angiogenic and antiangiogenic factors has emerged as a potential key pathway in the pathophysiology of preeclampsia. Patients with preeclampsia have a higher circulating concentration of antiangiogenic factors (ie, soluble vascular endothelial growth factor receptor-1 [sVEGFR- 1], also called soluble fms-like tyrosine kinase 1 [sFlt1]) and soluble endoglin (sEng)] and a lower maternal circulating concentration of free angiogenic factors (ie, vascular endothelial growth factor [VEGF] and placental growth factor [PlGF]) than patients with a normal pregnancy.

Bronchopulmonary dysplasia is the main respiratory sequelae of preterm birth. Its rate increased in preterm infants born from mother with preeclampsia. Recent studies showed that bronchopulmonary dysplasia is consistently accompanied by a reduction in the number of small arteries and on abnormal distribution of vessels within the distal lungs. This is associated with reduced lung VEGF expression. Infants with maternal preeclampsia had higher cord blood sFlt-1 but lower PlGF and VEGF circulating levels. There was a significantly positive relationship between birth weight and cord blood sFlt-1 levels, witness of consequences of these antiangiogenic factors on fetuses. However, no study to date has shown a correlation between the level of angiogenic and antiangiogenic factors and the main complications of preterm birth.

The main objective of this population-based study, ie in 24 intra uterine growth restricted preterm babies born before 30 weeks of gestational age from mother with preeclampsia, was to examine whether levels of sFlt1 at birth in maternal and umbilical cord blood and in the amniotic fluid is associated with an increased risk of BPD at 36 weeks of gestational age. The second objectives are to explore the link between the levels of angiogenic and antiangiogenic factors and the main complications of preterm birth, ie, necrotizing enterocolitis, intra-ventricular hemorrhage, periventricular leukomalacia or infection.

ELIGIBILITY:
Inclusion Criteria:

* Maternal preeclampsia
* Intra uterine growth restriction
* Preterm birth before 30 weeks of gestational age

Exclusion Criteria:

* Congenital malformation
* Eutrophic fetus
* Chorioamnionitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intra uterine growth restricted preterm babies born before 30 weeks of gestational age from mother with preeclampsia
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2012-06; Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Levels of sFlt1 (tyrosine kinase 1) at birth and the risk of bronchopulmonary dysplasia | at 36 weeks of gestational age
  The main objective of this population-based study, ie in 24 intra uterine growth restricted preterm babies born before 30 weeks of gestational age from mother with preeclampsia, was to examine whether levels of sFlt1 at birth in maternal and umbilical cord blood and in the amniotic fluid is associated with an increased risk of BPD at 36 weeks of gestational age.

SECONDARY OUTCOMES:
Levels of angiogenic and antiangiogenic factors at birth and the complications of preterm birth | at 36 weeks of gestational age
  The second objectives are to correlate the levels of angiogenic and antiangiogenic factors at birth, in maternal blood, cord blood and amniotic fluid, and the main complications of preterm birth, ie, necrotizing enterocolitis, intra-ventricular hemorrhage, periventricular leukomalacia or infection before 36 weeks of gestational age.

CONTACTS AND LOCATIONS:
Overall Officials: Elodie ZANA-TAIEB, MD, Principal Investigator — Hôpital Cochin
Locations (1):
- Cochin Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No